CLINICAL TRIAL: NCT01339806
Title: Phase IV Study of Cognitive Rehabilitation Effectiveness for Mild Traumatic Brain Injury
Brief Title: The Study of Cognitive Rehabilitation Effectiveness for Mild Traumatic Brain Injury
Acronym: SCORE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: The Defense and Veterans Brain Injury Center (U.S. Federal Agency); Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Principal Investigator, Amy Bowles, M.D., TBI Service Chief, Brooke Army Medical Center
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: C.2010.199
Record Dates: First submitted 2011-04-15; First posted 2011-04-21 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Traumatic Brain Injury With Brief Loss of Consciousness; Traumatic Brain Injury With No Loss of Consciousness
Keywords: mTBI; Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard of Care for mTBI Provider Arm (Other): Arm 1: Psychoeducational Control Group. Individuals assigned to arm 1 will receive psychoeducational materials specifically adapted for persistent management of symptoms and routine follow-up with medical providers (every three weeks). Additionally, subjects assigned to this group will receive medical care (e.g., psychopharmacological management of depression) and/or referral for symptom management (e.g., vestibular rehabilitation) of non-cognitive complaints, consistent with the current standard of care treatment model for managing post-concussive symptoms (see Figure below adapted with permission from authors; Brenner et al., 2009).
  Interventions: Behavioral: Informational Handout/Provider Visits
- Computer Based Therapy Group (Experimental): Arm 2: Non-therapist directed computerized cognitive rehabilitation. Individuals assigned to treatment arm 2 will receive ten hours of in-clinic, computerized treatment per week throughout the 6-week treatment trial. Participants will be scheduled for 2 hours per day, proctored by clinic staff (certified recreation therapist or neuropsychology technician) who will be responsible for recording daily performance, providing positive reinforcement of participation, and effort. Computer programs selected for this treatment trial include both skill-specific training (e.g., attention processes) and general cognitive activation. These computer programs are commercially available and advertised as "brain fitness" or "brain training."
  Interventions: Behavioral: Brainworks; Behavioral: Informational Handout/Provider Visits
- Cognitive Rehab Group (Experimental): Arm 3: Therapist-directed individualized cognitive rehabilitation. Individuals assigned to treatment arm 3 will receive 10 hours of individual and group cognitive rehabilitation treatment (including homework assignments) per week conducted by credentialed speech therapists and occupational therapists. The treatment components will include five hours of weekly individual therapy (one-hour sessions; two hours focused on compensatory strategies and three hours focused on restorative strategies), two hours of weekly group therapy (one hour sessions focused on compensatory strategies), and three hours of weekly computer-based "homework" proctored by clinic staff who will be responsible for recording performance, and providing positive reinforcement of participation and effort.
  Interventions: Behavioral: Cognitive Rehab; Behavioral: Informational Handout/Provider Visits
- Cognitive and Psychological Based Rehab (Experimental): Arm 4: Integrated interdisciplinary cognitive rehabilitation combined with cognitive-behavioral psychotherapy. Individuals assigned to treatment arm 4 will receive 10 hours of individual and group treatment per week conducted by credentialed therapists and doctoral-level psychologists. The treatment components will include four hours of weekly 1 hr individual therapy sessions; 2 hrs of cognitive rehabilitation, 1 hr of cognitive rehab & 1 hr of individual psychotherapy targeting anxiety/combat stress symptoms including relaxation training & exposure therapy and cognitive-behavioral principles, 3 hrs of weekly group therapy & three hours of weekly "homework" including 30-mins relaxation training, 30-mins cognitive-behavioral psychotherapy homework, and 2 hrs of computerized cognitive rehabilitation exercises proctored by clinic staff.
  Interventions: Behavioral: Cognitive Rehab; Behavioral: Informational Handout/Provider Visits

INTERVENTIONS:
Behavioral: Cognitive Rehab — APT-III, Other standard individual and group interventions.
  Other Names: APT-III
  Arms: Cognitive Rehab Group; Cognitive and Psychological Based Rehab
Behavioral: Brainworks — POSIT
  Other Names: POSIT
  Arms: Computer Based Therapy Group
Behavioral: Informational Handout/Provider Visits — Provider based visits every three weeks and informational handout given to patient in regulation with current standard of care procedures.

SUMMARY:
The objective of this trial is to evaluate the effectiveness of cognitive rehabilitation in OIF/OEF service members with a history of mild traumatic brain injury and persistent (3-24 months post injury) cognitive complaints. This is a prospective, randomized, control treatment trial of cognitive rehabilitation for OEF/OIF Service Members with a history of mild traumatic brain injury (mTBI) and persistent (3-24 months post-injury) cognitive complaints. Subjects will be recruited from consecutive patient referrals to the TBI Service at SAMMC-North. Patients who meet eligibility criteria and consent to participate in the treatment trial will be randomly assigned to one of four, 6-week treatment arms of the study. Subjects will be evaluated prior to the start of treatment and 3, 6, 12, and 18 weeks following the initiation of the study. The total number of patients to be studied is 160 (maximum), which is approximately 20 patients per month.

DETAILED DESCRIPTION:
This is a prospective, randomized, control treatment trial of cognitive rehabilitation for OEF/OIF Service Members with a history of mild traumatic brain injury (mTBI) and persistent (3-24 months post-injury) cognitive complaints. Subjects will be recruited from consecutive patient referrals to the TBI Service at SAMMC-North. Patients who meet eligibility criteria and consent to participate in the treatment trial will be randomly assigned to one of four, 6-week treatment arms of the study: 1. Psychoeducational control group; 2. Non-therapist directed, computerized cognitive rehabilitation; 3. Therapist-directed individualized cognitive rehabilitation; and 4. Integrated interdisciplinary cognitive rehabilitation combined with cognitive-behavioral psychotherapy. (Components of the treatment arms are described in detail in section 4.6; Research Design and Methods.) All subjects enrolled in the study will receive the standard of care in management of chronic post-concussive symptoms, consistent with the VA/DoD Clinical Practice Guidelines for the Management of Concussion/mild TBI (Barth et al., 2009), regardless of treatment assignment. The standard of care includes provision of patient education materials (adapted from existing studies to address more persistent rather than acute symptom management), regular scheduled follow-up with a medical provider every three weeks, and symptom-based treatment of post-concussive complaints (e.g., medication trials for headache and co-occurring psychiatric disorders, physical therapy for vestibular complaints, case management, and supportive counseling with social work for soldiers assigned to the Warriors-in-Transition Battalion). Study participants who are assigned to treatment arms 2, 3, or 4 will additionally receive manualized cognitive rehabilitation therapies during the 6-week treatment phase of the study. Cognitive rehabilitation treatment intensity (i.e., number of hours of treatment per week) will be matched for individuals assigned to treatment arms 2, 3, or 4. Participants assigned to the control treatment group (treatment arm 1) will be offered individualized cognitive rehabilitation therapy if their cognitive complaints do not abate following the completion of the six-week treatment trial.

Study participants will be evaluated prior to the initiation of treatment, as well as at 3-weeks, 6-weeks, 12-weeks, and 18-weeks following the start of treatment. Study evaluators will be blind to treatment assignment. Pre-treatment baseline assessments and peri-/post-treatment outcome assessments will include demographic information, injury-related variables, self-report inventories, performance on neuropsychological testing, and functional status (e.g., work status; healthcare utilization). Detailed descriptions of the data to be collected including primary and secondary outcome measures, as well as co-variate measures can be found in section 4.8: Instrumentation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mTBI as defined in the VA/DoD Clinical Practice Guidelines for the Management of Concussion/mild TBI (Barth et al., 2009) which occurred during deployment in support of OEF/OIF within 3-24 months of study enrollment;
* Presence of cognitive complaints (NSI score of 3 or higher on any of the four cognitive symptoms)
* Ability to understand and communicate in English.

Exclusion Criteria:

* Medical/psychiatric/neurologic co-morbidities of: blindness/low vision; uncontrolled seizure disorder; psychosis; history of moderate, severe TBI or penetrating BI; or Spinal Cord Injury with no use of upper extremities;
* Active participation in intensive (> 5 appointments per week) treatment for amputation, orthopedic trauma, burns, substance abuse, or post-traumatic stress disorder which would preclude full participation in an intensive cognitive rehabilitation program; or
* Daily use of narcotic pain medication(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2011-06; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Emotional Functioning | Baseline
  Symptom Checklist-90-Revised (SCL-90-R)
  Global Severity Index and 9 subscales:
  Somatization; Obsessive-Compulsive; Interpersonal Sensitivity; Depression; Anxiety; Hostility; Phobic Anxiety; Paranoid Ideation, and Psychoticism
Cognitive Efficiency | Baseline
  Paced Auditory Serial Addition Test (PASAT)
  * correct trial 1
  * correct trial 2
  * correct trial 3
  * correct trial 4 Sum of trials 1-4
Functional Behaviors | Baseline
  Key Behaviors Change Inventory (KBCI) Total score Inattention- raw & T-score Impulsivity- raw & T-score Unawareness of Problems - raw & T-score Apathy - raw & T-score Interpersonal Difficulties - raw & T-score Communication Problems - raw & T-score Somatic Difficulties - raw & T-score Emotional Adjustment - raw & T-score 64 individual items
Emotional Functioning | 3 Weeks
  Symptom Checklist-90-Revised (SCL-90-R)
  Global Severity Index and 9 subscales:
  Somatization; Obsessive-Compulsive; Interpersonal Sensitivity; Depression; Anxiety; Hostility; Phobic Anxiety; Paranoid Ideation, and Psychoticism
Emotional Functioning | 6 Weeks
  Symptom Checklist-90-Revised (SCL-90-R)
  Global Severity Index and 9 subscales:
  Somatization; Obsessive-Compulsive; Interpersonal Sensitivity; Depression; Anxiety; Hostility; Phobic Anxiety; Paranoid Ideation, and Psychoticism
Emotional Functioning | 12 Weeks
  Symptom Checklist-90-Revised (SCL-90-R)
  Global Severity Index and 9 subscales:
  Somatization; Obsessive-Compulsive; Interpersonal Sensitivity; Depression; Anxiety; Hostility; Phobic Anxiety; Paranoid Ideation, and Psychoticism
Emotional Functioning | 18 Weeks
  Symptom Checklist-90-Revised (SCL-90-R)
  Global Severity Index and 9 subscales:
  Somatization; Obsessive-Compulsive; Interpersonal Sensitivity; Depression; Anxiety; Hostility; Phobic Anxiety; Paranoid Ideation, and Psychoticism
Cognitive Efficiency | 3 Weeks
  Paced Auditory Serial Addition Test (PASAT)
  * correct trial 1
  * correct trial 2
  * correct trial 3
  * correct trial 4 Sum of trials 1-4
Cognitive Efficiency | 6 Weeks
  Paced Auditory Serial Addition Test (PASAT)
  * correct trial 1
  * correct trial 2
  * correct trial 3
  * correct trial 4 Sum of trials 1-4
Cognitive Efficiency | 12 Weeks
  Paced Auditory Serial Addition Test (PASAT)
  * correct trial 1
  * correct trial 2
  * correct trial 3
  * correct trial 4 Sum of trials 1-4
Cognitive Efficiency | 18 Weeks
  Paced Auditory Serial Addition Test (PASAT)
  * correct trial 1
  * correct trial 2
  * correct trial 3
  * correct trial 4 Sum of trials 1-4
Functional Behaviors | 3 Weeks
  Key Behaviors Change Inventory (KBCI) Total score Inattention- raw & T-score Impulsivity- raw & T-score Unawareness of Problems - raw & T-score Apathy - raw & T-score Interpersonal Difficulties - raw & T-score Communication Problems - raw & T-score Somatic Difficulties - raw & T-score Emotional Adjustment - raw & T-score 64 individual items
Functional Behaviors | 6 Weeks
  Key Behaviors Change Inventory (KBCI) Total score Inattention- raw & T-score Impulsivity- raw & T-score Unawareness of Problems - raw & T-score Apathy - raw & T-score Interpersonal Difficulties - raw & T-score Communication Problems - raw & T-score Somatic Difficulties - raw & T-score Emotional Adjustment - raw & T-score 64 individual items
Functional Behaviors | 12 Weeks
  Key Behaviors Change Inventory (KBCI) Total score Inattention- raw & T-score Impulsivity- raw & T-score Unawareness of Problems - raw & T-score Apathy - raw & T-score Interpersonal Difficulties - raw & T-score Communication Problems - raw & T-score Somatic Difficulties - raw & T-score Emotional Adjustment - raw & T-score 64 individual items
Functional Behaviors | 18 Weeks
  Key Behaviors Change Inventory (KBCI) Total score Inattention- raw & T-score Impulsivity- raw & T-score Unawareness of Problems - raw & T-score Apathy - raw & T-score Interpersonal Difficulties - raw & T-score Communication Problems - raw & T-score Somatic Difficulties - raw & T-score Emotional Adjustment - raw & T-score 64 individual items

SECONDARY OUTCOMES:
Fatigue | Baseline
  Fatigue Severity Scale (FSS) Total Raw scale 9 individual items
Post-Concussive Symptoms | Baseline
  Neurobehavioral Symptom Inventory Total Raw scale 22 individual items
Self Reported Quality of Life | Baseline
  World Health Organization Brief Quality of Life Scale (WHO-QOL-BREF) Total transformed score
  Total score for each of the 5 subscale domains:
  Overall Functioning Physical Capacity Psychological Social Relationships Environment
Neuropsychological Status | Baseline
  Neuropsychological Global Composite Score Average normative t-score of: [CVLT-2 sum trials 1-5, D-KEFS Verbal Fluency total score, Trail Making Test - part B only, WAIS-IV Processing Speed, Working, CVLT- 2 Trial 1, CVLT-2 Trial 2, CVLT- 2 Trial 3, CVLT-2 Trial 4, CVLT-2 Trial 5, CVLT-2 Total Trials 1-5, CVLT-2 Total Trials 1-5 (T-score), CVLT-2 List B, SDFR, SDCR, LDFR, LDCR, total perseverations,total intrusions CVLT-2 LD recognition hits CVLT-2 LD recognition FP errors Trails part A, Trails part B, Trails part A, Trails part B, WAIS-IV Processing Speed Index, WAIS-IV Symbol Search
Self Reported Alcohol Use Behaviors | Baseline
  Alcohol Use Disorders Identification Test (AUDIT) Summary Socre; 10 individual items
Post-Traumatic Stress Symptomatology | 18 Weeks
  Post-Traumatic Stress Checklist-Military Form (PCL-M) Total Raw Socre 17 items
Self Reported Headache Disability | Baseline
  Headache Impact Test-6 (HIT-6) Total Weighted Score
Health Related (Cognition) Locus of Control | Baseline
  Multidimensional Health Locus of Control Scale (MHLCS-Form C) Internal subscale-total raw Chance subscale-total raw Powerful others subscale-total raw Doctors subscale-total raw Other people subscale-total raw
Perceived Self-Efficacy (Cognition) | Baseline
  Self-Efficacy for Symptom Management Scale SEsx total SEsocial subscale SEemotional subscale SEcognitvie subscale 13 individual items
Attribution of Cognitive Symptoms | Baseline
  Cognitive Symptom Attribution Scale 7 individual items
Therapist-Rated Patient Engagement in Treatment | Week 6 of treatment
  Rehabilitation Intensity of Therapy Scale (RITS) Weekly average rating (weeks 1-6)
Post-Concussive Symptoms | 6 Weeks
  Neurobehavioral Symptom Inventory (NSI) Total Raw scale 22 individual items
Post-Concussive Symptoms | 12 weeks
  Neurobehavioral Symptom Inventory (NSI) Total Raw scale 22 individual items
Post-Concussive Symptoms | 18 weeks
  Neurobehavioral Symptom Inventory (NSI) Total Raw scale 22 individual items
Fatigue | 6 weeks
  Fatigue Severity Scale (FSS) Total Raw scale 9 individual items
Fatigue | 12 Weeks
  Fatigue Severity Scale (FSS) Total Raw scale 9 individual items
Fatigue | 18 Weeks
  Fatigue Severity Scale (FSS) Total Raw scale 9 individual items
Change in Healthcare Utilization | 30 days prior to Baseline and 6 months post Baseline
  Summed total number of appointments 30 days prior to study enrollment and summed total number of appointments for 30 days between 5 and 6 months post-treatment.
Self Reported Quality of Life | 6 weeks
  World Health Organization Brief Quality of Life Scale (WHO-QOL-BREF) Total transformed score
  Total score for each of the 5 subscale domains:
  Overall Functioning Physical Capacity Psychological Social Relationships Environment
Self Reported Quality of Life | 12 weeks
  World Health Organization Brief Quality of Life Scale (WHO-QOL-BREF) Total transformed score
  Total score for each of the 5 subscale domains:
  Overall Functioning Physical Capacity Psychological Social Relationships Environment
Self Reported Quality of Life | 18 weeks
  World Health Organization Brief Quality of Life Scale (WHO-QOL-BREF) Total transformed score
  Total score for each of the 5 subscale domains:
  Overall Functioning Physical Capacity Psychological Social Relationships Environment
Neuropsychological Status | 6 Weeks
  Neuropsychological Global Composite Score Average normative t-score of: [CVLT-2 sum trials 1-5, D-KEFS Verbal Fluency total score, Trail Making Test - part B only, WAIS-IV Processing Speed, Working, CVLT- 2 Trial 1, CVLT-2 Trial 2, CVLT- 2 Trial 3, CVLT-2 Trial 4, CVLT-2 Trial 5, CVLT-2 Total Trials 1-5, CVLT-2 Total Trials 1-5 (T-score), CVLT-2 List B, SDFR, SDCR, LDFR, LDCR, total perseverations,total intrusions CVLT-2 LD recognition hits CVLT-2 LD recognition FP errors Trails part A, Trails part B, Trails part A, Trails part B, WAIS-IV Processing Speed Index, WAIS-IV Symbol Search
Neuropsychological Status | 12 Weeks
  Neuropsychological Global Composite Score Average normative t-score of: [CVLT-2 sum trials 1-5, D-KEFS Verbal Fluency total score, Trail Making Test - part B only, WAIS-IV Processing Speed, Working, CVLT- 2 Trial 1, CVLT-2 Trial 2, CVLT- 2 Trial 3, CVLT-2 Trial 4, CVLT-2 Trial 5, CVLT-2 Total Trials 1-5, CVLT-2 Total Trials 1-5 (T-score), CVLT-2 List B, SDFR, SDCR, LDFR, LDCR, total perseverations,total intrusions CVLT-2 LD recognition hits CVLT-2 LD recognition FP errors Trails part A, Trails part B, Trails part A, Trails part B, WAIS-IV Processing Speed Index, WAIS-IV Symbol Search
Neuropsychological Status | 18 Weeks
  Neuropsychological Global Composite Score Average normative t-score of: [CVLT-2 sum trials 1-5, D-KEFS Verbal Fluency total score, Trail Making Test - part B only, WAIS-IV Processing Speed, Working, CVLT- 2 Trial 1, CVLT-2 Trial 2, CVLT- 2 Trial 3, CVLT-2 Trial 4, CVLT-2 Trial 5, CVLT-2 Total Trials 1-5, CVLT-2 Total Trials 1-5 (T-score), CVLT-2 List B, SDFR, SDCR, LDFR, LDCR, total perseverations,total intrusions CVLT-2 LD recognition hits CVLT-2 LD recognition FP errors Trails part A, Trails part B, Trails part A, Trails part B, WAIS-IV Processing Speed Index, WAIS-IV Symbol Search
Self Reported Alcohol Use Behaviors | 6 weeks
  Alcohol Use Disorders Identification Test (AUDIT) Summary Socre; 10 individual items
Self Reported Alcohol Use Behaviors | 12 weeks
  Alcohol Use Disorders Identification Test (AUDIT) Summary Socre; 10 individual items
Self Reported Alcohol Use Behaviors | 18 weeks
  Alcohol Use Disorders Identification Test (AUDIT) Summary Socre; 10 individual items
Post-Traumatic Stress Symptomatology | 6 weeks
  Post-Traumatic Stress Checklist-Military Form (PCL-M) Total Raw Socre 17 items
Post-Traumatic Stress Symptomatology | Baseline
  Post-Traumatic Stress Checkilist-Military Form (PCL-M) Total Raw Socre 17 items
Post-Traumatic Stress Symptomatology | 12 Weeks
  Post-Traumatic Stress Checklist-Military Form (PCL-M) Total Raw Socre 17 items
Self Reported Headache Disability | 6 weeks
  Headache Impact Test-6 (HIT-6) Total Weighted Score
Self Reported Headache Disability | 12 weeks
  Headache Impact Test-6 (HIT-6) Total Weighted Score
Self Reported Headache Disability | 18 Weeks
  Headache Impact Test-6 (HIT-6) Total Weighted Score
Health Related (Cognition) Locus of Control | 6 weeks
  Multidimensional Health Locus of Control Scale (MHLCS-Form C) Internal subscale-total raw Chance subscale-total raw Powerful others subscale-total raw Doctors subscale-total raw Other people subscale-total raw
Health Related (Cognition) Locus of Control | 12 weeks
  Multidimensional Health Locus of Control Scale (MHLCS-Form C) Internal subscale-total raw Chance subscale-total raw Powerful others subscale-total raw Doctors subscale-total raw Other people subscale-total raw
Health Related (Cognition) Locus of Control | 18 weeks
  Multidimensional Health Locus of Control Scale (MHLCS-Form C) Internal subscale-total raw Chance subscale-total raw Powerful others subscale-total raw Doctors subscale-total raw Other people subscale-total raw
Perceived Self-Efficacy (Cognition) | 6 weeks
  Self-Efficacy for Symptom Management Scale SEsx total SEsocial subscale SEemotional subscale SEcognitvie subscale 13 individual items
Perceived Self-Efficacy (Cognition) | 12 weeks
  Self-Efficacy for Symptom Management Scale SEsx total SEsocial subscale SEemotional subscale SEcognitvie subscale 13 individual items
Perceived Self-Efficacy (Cognition) | 18 weeks
  Self-Efficacy for Symptom Management Scale SEsx total SEsocial subscale SEemotional subscale SEcognitvie subscale 13 individual items
Attribution of Cognitive Symptoms | 6 weeks
  Cognitive Symptom Attribution Scale 7 individual items
Attribution of Cognitive Symptoms | 12 weeks
  Cognitive Symptom Attribution Scale 7 individual items
Attribution of Cognitive Symptoms | 18 weeks
  Cognitive Symptom Attribution Scale 7 individual items
Therapist-Rated Patient Engagement in Treatment | Week 1 of Treatment
  Rehabilitation Intensity of Therapy Scale (RITS) Weekly average rating (weeks 1-6)
Therapist-Rated Patient Engagement in Treatment | Week 2 of treatment
  Rehabilitation Intensity of Therapy Scale (RITS) Weekly average rating (weeks 1-6)
Therapist-Rated Patient Engagement in Treatment | Week 3 of treatment
  Rehabilitation Intensity of Therapy Scale (RITS) Weekly average rating (weeks 1-6)
Therapist-Rated Patient Engagement in Treatment | Week 4 of treatment
  Rehabilitation Intensity of Therapy Scale (RITS) Weekly average rating (weeks 1-6)
Therapist-Rated Patient Engagement in Treatment | Week 5 of treatment
  Rehabilitation Intensity of Therapy Scale (RITS) Weekly average rating (weeks 1-6)

CONTACTS AND LOCATIONS:
Overall Officials: Amy O Bowles, MD, Principal Investigator — BAMC
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

REFERENCES:
- [Derived] Vanderploeg RD, Cooper DB, Curtiss G, Kennedy JE, Tate DF, Bowles AO. Predicting treatment response to cognitive rehabilitation in military service members with mild traumatic brain injury. Rehabil Psychol. 2018 May;63(2):194-204. doi: 10.1037/rep0000215. PMID 29878826
- [Derived] Cooper DB, Bowles AO, Kennedy JE, Curtiss G, French LM, Tate DF, Vanderploeg RD. Cognitive Rehabilitation for Military Service Members With Mild Traumatic Brain Injury: A Randomized Clinical Trial. J Head Trauma Rehabil. 2017 May/Jun;32(3):E1-E15. doi: 10.1097/HTR.0000000000000254. PMID 27603763
- See also: Defense and Veterans Brain Injury Center — http://www.dvbic.org/